CLINICAL TRIAL: NCT02546076
Title: Within-subject Randomized Clinical Trial Comparing Dual-mode ER:YAG Laser in Patients With Long Keloid/Hypertrophic Scars
Brief Title: Comparison of Dual-mode ER:YAG Laser in Patients With Long Keloid/Hypertrophic Scars
Acronym: KELOID
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of patients
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KELOID
Record Dates: First submitted 2015-09-02; First posted 2015-09-10 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Keloid; Hypertrophic Scars
Keywords: Keloid; Hypertrophic scars; Er-YAG Lasers
MeSH Terms: conditions — Keloid; Cicatrix, Hypertrophic | interventions — Laser Coagulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laser coagulation (Active Comparator): Er:YAG laser treatment with coagulation modality
  Interventions: Device: Laser coagulation
- Laser w/o coagulation (Active Comparator): Er:YAG laser treatment without coagulation modality
  Interventions: Device: Laser w/o coagulation

INTERVENTIONS:
Device: Laser coagulation — The treatment consists in performing Er:Yag laser with long-pulsed Erbium mode
  Arms: Laser coagulation
Device: Laser w/o coagulation — The treatment consists in performing Er:Yag laser with true pulsed Erbium mode
  Arms: Laser w/o coagulation

SUMMARY:
Skin injuries due to trauma are relatively common, and patients are very concerned about scars caused by trauma and primary repair. Recently, the use of ablative and non-ablative lasers based on the fractional approach has become a novel strategy for the treatment of scars.

The objective of this study is to compare the efficacy of dual-mode Er:YAG laser delivering pulses either with and without heat/coagulation in a cohort of patients with long keloid/hypertrophic scars.

The main hypothesis is that ablative fractional laser without heat/coagulation is equivalent to laser with heat/coagulation in terms of scars volume reduction, while the secondary hypothesis is that ablative fractional laser without heat/coagulation is superior in terms of post-operative erythema and hypopigmentation reduction.

DETAILED DESCRIPTION:
Background

Skin injuries, such as lacerations or abrasions, due to trauma are relatively common, and patients are very concerned about scars caused by trauma and primary repair. Multiple modalities for improving the clinical appearance of scars have been attempted with varying success, including corticosteroids, dermabrasion, surgical revision, chemical peeling, silicone gel application, pressure therapy, and radiation. Lasers such as the carbon dioxide (CO2), erbium: yttrium-aluminum-garnet (Er:YAG), and pulsed dye (PDL) lasers have all been used with differing success in the treatment of scars. The goal of all these treatments is to soften depressions and stimulate neocollagenesis in order to fill in the residual defects.

Ablative lasers used for skin resurfacing, such as the CO2 and Er:YAG laser, can reduce various scars, but significant adverse effects limit their use, and patient downtime can be extensive. Owing to these potential risks, nonablative lasers have been developed as a safe alternative to ablative laser resurfacing, and have been reported to be effective and safe for scars. However outcomes have remained unsatisfactory and require several treatments to achieve satisfactory efficacy.

Recently, the use of ablative and non-ablative lasers based on the fractional approach has become a novel strategy for the treatment of scars, and some authors have suggested that treatment with fractional lasers for various scars, such as postoperative, atrophic, and acne scars, has been demonstrated to safely improve the appearance of the scars. However, there is a lack of studies comparing coagulation modality of such lasers.

Objective

The objective of this study is to compare the efficacy of dual-mode Er:YAG laser delivering pulses either with and without heat/coagulation in a cohort of patients with long keloid/hypertrophic scars.

Methods

This is a single center, investigator initiated, double blind, within-subject split-lesion design, equivalence randomized clinical study.

Consecutive patients, referring to Dermatology outpatient and fulfilling inclusion criteria, are included. Participants are then randomly assigned to get treatment with Er:YAG laser on half of scar section side by equally splitting the lesion area in two symmetric and uniform parts. One side will be treated with coagulation while the other one will be without. In case of multiple lesions per patient, only the largest and most uniform one is selected for the study purpose.

ELIGIBILITY:
Inclusion Criteria:

* Given written informed consent
* Skin type I-IV
* Presence of long keloid/hypertrophic scar of at least 3 cm² and of uniform/symmetric type
* Willingness and ability to adhere study protocol

Exclusion Criteria

* History of adverse events related to ablative fractional laser therapy
* Ablative resurfacing within the last 6 months on the scar
* Oral retinoid, any immunosuppressive treatments in the last 6 months
* Pregnancy, lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Any reduction from baseline of scars volume as assessed by image analysis | 24 weeks

SECONDARY OUTCOMES:
Any reduction from baseline of scars volume as assessed by image analysis | 4, 8, 12, 16, 24 weeks
Any improvement of scars as assessed by physician according to an ordinal 6-points scale | 4, 8, 12, 16, 24 weeks
Overall patient satisfaction to the proposed therapy as assessed by visual analogue scale | 16, 24 weeks
Erythema index as assessed by image analysis | 4, 8, 12, 16, 24 weeks
Hypopigmentation as assessed by image analysis | 4, 8, 12, 16, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Adatto, MD, Principal Investigator — Dep. of Dermatology, Inselspital University Hospital, Bern (Switzerland)